CLINICAL TRIAL: NCT03698747
Title: A Prospective Study of Myelin Imaging Changes in Concussed High School Football Players
Brief Title: Myelin Imaging in Concussed High School Football Players
Status: Terminated | Type: Observational
Why Stopped: PI left organization
Sponsor: Memorial Healthcare System (Other)
Responsible Party: Sponsor
Other Study IDs: MTBI
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- mTBI Study Group with McDESPOT sequence: Study group (30 subjects) of football players diagnosed with mTBI (scan at diagnosis, 3-month follow-up scan, genetic screening, concussion assessment at both interaction)
  Interventions: Device: McDESPOT
- Control Group: Control group (30 subjects) of age match non-contact sport players (scan, genetic testing, concussion assessment)

INTERVENTIONS:
Device: McDESPOT — myelin specific MRI sequence (mcDESPOT) added to standard MRI sequence
  Groups: mTBI Study Group with McDESPOT sequence

SUMMARY:
Investigate myelin alterations in high school football players with mTBI

DETAILED DESCRIPTION:
The lack of highly sensitive clinical neuroimaging and neuropsychiatric markers of subtle changes due to mTBI makes it difficult to characterize injury severity and to predict outcomes. White matter tracts in the brain, both myelinated and non-myelinated, are susceptible to damage from impact-acceleration forces experienced during a TBI,5-7 and there is evidence that significant white matter injury and myelin loss occurs in mTBI. In addition, this damage may be chronic and can negatively affect neural processing speed and cognitive function. Traditional anatomical and function MRI imaging sequences include clinical sequences such as traditional T1 and T2 sequences, fluid-attenuated inversion recovery (FLAIR), three-dimensional (3D) magnetization-prepared rapid gradient echo (MP-RAGE), diffusion-weighted imaging (DWI) and gradient MRI. While a number of advanced imaging techniques, notably magnetization transfer, diffusion tensor and quantitative T1 and T2 imaging (MTI, DTI, qT1 and qT2, respectively), have been used previously to study white matter in neurosurgical diseases, these methods provide only indirect, non-specific information related to myelin content. For example, these modalities can tell when there is swelling that is affecting the movement of water, which may be indicative of a process that would affect myelin, but they cannot give specific information about the amount of myelin surrounding a nerve. An emerging multicomponent relaxometry technique, termed multicomponent driven equilibrium single pulse observation of T1 and T2 (mcDESPOT), provides a voxel-wise estimation ranging from 0 to 1 for myelin content, with higher values providing an indirect marker of greater myelin integrity. Two studies have shown increased myelin after injury in football and ice hockey players.8 DTI, which primarily gives information about the myelin-axon bundle interactions, has shown decreased fractional anisotropy after mTBI,myelin-axon bundle interactions, has shown decreased fractional anisotropy after mTBI, indicating that the myelin that is present is less organized.8 Combining mcDESPOT and DTI findings, it is possible to see a more nuanced picture of the remyelination process after mTBI. In the present program, the investigators propose adding the mcDESPOT sequence to the MRI scanner in accordance with the MRI manufacturer's technical requirements. Although the sequences obtained for mcDESPOT are nearly identical sequences used in clinical practice, the flip-angles are changed so that they cannot be read like a traditional image.

Rather, the data have to be post-processed by a computer in order to be able to derive myelin information. The mcDESPOT sequences are FDA approved, and present no additional risk over traditional clinical MRI sequences. Apolipoprotein E (ApoE) is a class of proteins involved in the metabolism of fats in the body, and is important in Alzheimer's disease and cardiovascular disease. How the body makes this protein is genetically coded in the APoE gene. One form of this gene, APoE allele 4 (APoE4) is found in about 25% of the population, but in 60% of patients with Alzheimer's dementia. Infants with this allele also show decreased myelination at a young age. It is postulated that this defect affects the brain's ability to myelinate and remyelinate, leading to decreased or disorganized myelination, which then leads to an increased risk for development of dementia. This study aims to build upon preliminary data collected by the principal investigator (PI) showing increased but disorganized myelin in collegiate football players, by confirming and reproducing these results in a larger population. This study will also add the component of genetic testing for the APoE4 allele to see if there is a sub-segment of the study population that may be at increased risk for brain injury after mTBI and subsequent findings in the research scans. The mcDESPOT and genetic testing findings will also be correlated with routine neuropsychology concussion assessment results.

ELIGIBILITY:
Inclusion Criteria:

* Experimental Group

  * Patient age range: 9th through 12th grade (high school)
  * Male
  * Right-handed
  * Diagnosis of mTBI or concussion during a football game or training
  * No significant co-morbidities
  * Able to get an MRI
  * Potential subject must be capable of giving informed consent or assent when applicable

    • Control Group
  * Patient age range: 9th through 12th grade (high school)
  * Male Right-handed
  * Does not play contact sports (football, soccer, lacrosse)
  * No significant co-morbidities
  * Able to get an MRI
  * Potential subject must be capable of giving informed consent or assent when applicable

Exclusion Criteria:

* Unable to tolerate MRI scan

Ages: 13 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes — Male high school football players
Study Population: High school age (9th-12th grade), male, right-handed Diagnosed with concussion or mild traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Myelin Disruption on MRI brain scan | 3 months
  Determine whether mTBI in football players leads to increased, but disorganized, myelin compared to non-contact sports players.

SECONDARY OUTCOMES:
APoE4 allele genetic mutation on blood test | 3 months
  Explore whether a genetic mutation in the APoE4 allele predisposes football players to decreased or disorganized myelination after mTBI.
Neuropsychiatric concussion correlation | 3 months
  Correlate any changes in myelination or of genetics with neuropsychiatric concussion assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Spader, MD, Principal Investigator — Memorial Healthcare System
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No